CLINICAL TRIAL: NCT00453414
Title: Safety and Efficacy of Inhaled Iloprost in Pediatric Patients With Pulmonary Arterial Hypertension
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to lack of enrollment
Sponsor: Actelion (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C200-007
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; Pediatric; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Iloprost

INTERVENTIONS:
Drug: Iloprost Inhalation Solution (Ventavis)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of iloprost for PAH in children who are between the ages of 3 and 18 years old.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 3-18 years
* Diagnosis of PAH due to IPAH, connective tissue disease, or congenital heart disease
* Pulmonary arterial hypertension confirmed by a cardiac catheterization, with mPAP > 25 mmHg at rest, PCWP or LVEDP ≤ 15 mmHg, and PVR ≥ 240 dynes/sec/cm-5 (ie, ≥ 3.0 units m2)
* NYHA/WHO functional Class II, III, or IV
* Have had a 6-minute walk test (6-MWT) performed within the 3 months preceding the screening visit (if ≥ 8 years of age)
* Have had cardiopulmonary exercise testing (CPET) performed within the 3 months preceding the screening visit (if ≥ 8 years of age and > 130 cms in height. CPET testing will be conducted on NYHA/WHO Class IV patients at the discretion of the Principal Investigator)
* If receiving therapy for PAH, on a stable dose and regimen for at least 3 months prior to the screening visit
* If receiving digoxin, diuretic, or oxygen therapy, on a stable dose and regimen for at least 30 days preceding the screening visit
* Must demonstrate the ability to appropriately use the nebulizer device as part of the screening process

Exclusion Criteria:

* Prior use of prostacyclins or prostacyclin analogues within 3 months prior to screening
* Portal hypertension or clinically relevant hepatic disease
* Eisenmenger syndrome with resting SpO2 <88% on room air
* Clinically relevant asthma or other chronic lung disease, such as bronchopulmonary dysplasia, cystic fibrosis, or repaired or unrepaired congenital diaphragmatic hernia
* Diagnosis or current evidence of active lung infection or clinically relevant hemoptysis
* Left-sided heart disease, including valvular disease or heart failure
* Initiation or dosage adjustment of PAH-specific therapy within 3 months prior to screening
* Initiation of treatment with digoxin, diuretics, anticoagulation, or oxygen therapy within 30 days prior to screening

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07; Primary Completion 2006-10 (Estimated); Study Completion 2006-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 6-minute walk distance measured post-inhalation (for patients ≥ 8 years old) at Week 8 and Week 16
Change from baseline in Borg Dyspnea Scale measured following 6-MWT (for patients ≥ 8 years old) at Week 8 and Week 16
Change from baseline in NYHA/WHO functional class at Week 8 and Week 16
Change from baseline in hemodynamic parameters measured at Week 16, and in patients who are able to undergo iloprost inhalation while consciously sedated, hemodynamic parameters measured prior to dosing and 15-30 minutes after dosing
Time to clinical worsening, defined as any one of the following: death due to underlying PAH, transplantation, atrial septostomy, hospitalization for PAH or right heart failure, >15% worsening in 6-minute walk distance in concert with a ≥ 1 class deteri
Change from baseline in Child Health Questionnaire (CHQ-28) at Week 8 and Week 16
Change from baseline in exercise capacity, as measured by post-inhalation CPET, at Week 8 and Week 16 (if ≥ 8 years old and > 130 cms in height. CPET testing will be conducted on NYHA/WHO Class IV patients at the discretion of the Principal Investigat

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Children's Hospital, Denver, Colorado
  - Columbia University Medical Center, New York, New York